CLINICAL TRIAL: NCT01086618
Title: A Randomized Trial of Initial Surgery in Advanced Asymptomatic Colorectal Cancer Patients Receiving Chemotherapy for Metastatic Disease
Brief Title: Chemotherapy With or Without Surgery in Treating Patients With Metastatic Colorectal Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University College London Hospitals (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000667364; UCL-08/0079; UCL-ISAAC; ISRCTN10963271; EU-21008; CRUK-C32436/A10431; EUDRACT-2008-005911-16; MREC-09/H1102/60; NCRI-UCL-08/0079
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2010-03

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Neoadjuvant Therapy; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: systemic chemotherapy
Procedure: adjuvant therapy
Procedure: quality-of-life assessment
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy after surgery may kill any tumor cells that remain after surgery. It is not yet known whether chemotherapy is more effective when given alone or together with surgery in treating patients with colorectal cancer.

PURPOSE: This randomized phase II/III trial is studying how well chemotherapy works and compares it with surgery followed by chemotherapy in treating patients with metastatic colorectal cancer that can not be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine whether overall survival is improved in patients with asymptomatic, unresectable metastatic colorectal cancer treated with chemotherapy alone versus surgery followed by chemotherapy.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I (control arm): Patients receive systemic chemotherapy according to standard local practice. Patients who develop symptoms from their primary tumor receive treatment as required including surgery, if indicated.
* Arm II (experimental arm): Patients undergo surgery at the discretion of the surgeon. Beginning 8 weeks after completion of surgery, patients receive chemotherapy according to standard local practice.

Patients complete quality-of-life questionnaires (EQ-5D) at baseline and then periodically during and after completion of study treatment.

After completion of study treatment, patients are followed every 3 months.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed colorectal cancer

  * Metastases which are unresectable at presentation
* No known unresectable primary tumor on CT/MRI scan
* Primary tumor does not require immediate or emergency intervention including surgery, radiotherapy, laser, or stenting

  * Patients who are treated with colonic stents are eligible
* No unequivocal extensive peritoneal metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Must be fit for systemic chemotherapy and surgery
* Hemoglobin > 10.0 g/dL
* WBC > 3.0 x 10^9/L
* Platelet count > 100 x 10^9/L
* Bilirubin < 25 μmol/L
* GFR > 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months (female) or up to 2 months (male) after completion of study therapy
* No history of malignant disease within the past 5 years except for nonmelanomatous skin cancer or carcinoma in situ of the cervix
* No serious medical co-morbidity (e.g., uncontrolled inflammatory bowel disease, uncontrolled angina, recent [within the past 6 months] myocardial infarction, or another serious medical condition) judged to compromise ability to tolerate chemotherapy and/or surgery

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Concurrent participation in a trial of chemotherapy, if eligible, allowed
* Concurrent short-course radiotherapy for operable rectal cancer allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Accrual rate in months 10 to 12 (phase II)
Overall survival for ≥ 2 years (phase III)

SECONDARY OUTCOMES:
Morbidity of surgery (phase II)
Percentage of patients who receive chemotherapy following surgery (must be over 80%) (phase II)
Morbidity of chemotherapy and surgery (phase III)
Quality of life (phase III)
Economic evaluation (phase III)

CONTACTS AND LOCATIONS:
Overall Officials: Austin Obichere, MD, Principal Investigator — University College London Hospitals
Locations (1):
- University College Hospital, London, England, United Kingdom